CLINICAL TRIAL: NCT01089322
Title: Risk Factors Associated to Difficult-to-control Asthma: Characterization of Clinical, Structural and Inflammatory Factors Related to Treatment Response
Brief Title: Risk Factors Associated to Difficult-to-control Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rafael Stelmach (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Rafael Stelmach, MD-PHD, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBSTRUÇÃOHC-02
Record Dates: First submitted 2010-02-22; First posted 2010-03-18 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: ASTHMA
Keywords: SEVERE ASTHMA; RISK FACTORS; CHARACTERIZATION; CLINICAL CONTROL; INFLAMMATORY MARKERS; SEVERE; CONTROL
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Retrospective analysis after treatment outcome (controlled vs. non controlled) based on the primary outcome; and post hoc analysis after oral steroid treatment based on pulmonary function reversibility
Masking Description: Open label study. All subjects received the same treatment
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stantardized treament (Experimental): oral and inhaled corticosteroid plus LABA
  Interventions: Drug: inhaled corticosteroid plus LABA plus oral corticosteroid

INTERVENTIONS:
Drug: inhaled corticosteroid plus LABA plus oral corticosteroid — formoterol plus budesonide 12/400mcg 2times/day and 6/200 mcg as needed and prednisone 40 mcg
  Other Names: inhaled corticosteroid; LABA; oral corticosteroid

SUMMARY:
Several studies have demonstrated the efficacy of asthma treatment but despite being correctly diagnosed, conveniently prescribed and adherent to the therapeutics, 5% to 10% of asthmatics do not reach disease control.

The aim of this study is to measure asthma control, evaluate inflammatory and functional characteristics, describe comorbidities and aggravating factors and phenotypes derived from the characteristics of a severe asthmatic population followed at an outpatient university service in Sao Paolo, Brazil.

DETAILED DESCRIPTION:
Study design: interventional

Patients selection:

Seventy-four severe asthma patients, aged between 18 and 65 years old were recruited from the outpatient clinics of the Pulmonary Division of the University of São Paolo Hospital.

Severe asthma were defined according to GINA. Intervention: after 2 weeks screening period patients were treated with high inhaled corticosteroid dose plus long acting beta 2 agonist during 12 weeks plus oral corticosteroid ( prednisone 40 mg/day) during 2 weeks.

Procedures ( baseline, after 2 weeks and 12 weeks): asthma control questionnaire (ACQ), asthma control (ACT) test, lung function test, quality of life questionnaire (SGRQ and SF-36), exhaled nitric oxide (FeNO), induced sputum (IS). After 12 weeks patients underwent the following evaluation: Upper Digestive Endoscopy, Esophageal 24hs pHmetry, High Resolution Chest Tomography, Nasoscope exam,Bronchofibroscopy with endobronchial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of moderate to severe asthma (GINA) for at least one year
* Presence of airway obstruction reversibility (documented within the last 5 years before the start-up of study)
* Smoking, non-smoking or ex-smoking patients of <30 pack-years.
* Need of inhaled corticosteroid (IC),> or equal 1000mcg of Beclomethasone Dipropionate (DPB) or similar in the last year plus beta 2 long duration agonist in the last year.
* At least one exacerbation with the need of oral corticosteroid in the last year.

Exclusion Criteria:

* Pregnant women;
* Co-morbidities that may interfere with the management of the study;
* Patients who cannot understand the procedures of the study or who are not able to provide their free and clarified consent;
* Patients with other pulmonary diseases which may interfere with the evaluation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-12-09 (Actual); Primary Completion 2009-04-03 (Actual); Study Completion 2009-05-13 (Actual)

PRIMARY OUTCOMES:
Asthma control questionnaire (ACQ) | Baseline, after 2 weeks of oral corticosteroid trial and after 12 weeks of inhaled corticosteroid plus LABA
  Compare ACQ score in baseline and after 2 weeks of oral plus inhaled corticosteroid plus LABA and after 12 weeks of inhaled corticosteroid plus LABA

SECONDARY OUTCOMES:
Inflammatory parameters | Baseline, after 2 weeks of oral corticosteroid trial and after 12 weeks of inhaled corticosteroid plus LABA
  Compare inflammatory parameters ( FeNO and Induced sputum) at baseline and after 2 weeks of oral plus inhaled corticosteroid plus LABA and after 12 weeks of inhaled corticosteroid plus LABA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Regina M. Carvalho Pinto, MD, Principal Investigator — Heart Institute, University of São Paulo; Rafael Stelmach, PhD, Study Director — Heart Institute, University of São Paulo
Locations (1):
- University of São Paulo - Heart Institute and Hospital das Clínicas, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Athanazio R, Carvalho-Pinto R, Fernandes FL, Rached S, Rabe K, Cukier A, Stelmach R. Can severe asthmatic patients achieve asthma control? A systematic approach in patients with difficult to control asthma followed in a specialized clinic. BMC Pulm Med. 2016 Nov 16;16(1):153. doi: 10.1186/s12890-016-0314-1. PMID 27852260
- [Derived] de Carvalho-Pinto RM, Cukier A, Angelini L, Antonangelo L, Mauad T, Dolhnikoff M, Rabe KF, Stelmach R. Clinical characteristics and possible phenotypes of an adult severe asthma population. Respir Med. 2012 Jan;106(1):47-56. doi: 10.1016/j.rmed.2011.08.013. Epub 2011 Sep 3. PMID 21890336